CLINICAL TRIAL: NCT01770821
Title: REHABILITATION AFTER INTENSIVE CARE What Effect Does Physiotherapy and Proteinrich Sip Drink Have on Physical Performance, Bodycomposition, Bodyweight and Quality of Life?
Brief Title: Rehabilitation After Intensive Care
Acronym: REHAB
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of resource
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2009-2134; Innovest (Other: Haukeland University Hospital)
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Rehabilitation of Muscle Strength
Keywords: sip drink; protein; muscle strength; 6 minutes walking test

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standard physical training & standard nutrition (Active Comparator): Standard of care
  Interventions: Other: Dietary supplement and/or physical training
- Tailored physical training and sipdrink (Experimental): Tailored physical training and sipdrink (Protein nutridrink, 200 ml x 2)
  Interventions: Other: Dietary supplement and/or physical training
- Tailored physical training and standard nutrition. (Experimental): Standard physical training provided by the hospital and standard hospital nutrition
  Interventions: Other: Dietary supplement and/or physical training
- Standard physical training and sip drink (Experimental): Standard physical training provided by the hospital and sipdrink (Nutridrink protein, 200 ml x2)
  Interventions: Other: Dietary supplement and/or physical training

INTERVENTIONS:
Other: Dietary supplement and/or physical training

SUMMARY:
Patients with critical illness loose bodymass, mainly muscle. The purpose of the present study is to evaluate wheather tailored physical training and/or a sip drink (proteinrich) have effect on the six minutes walking test (6MWT), muscle strength, body weight, body composition and quality of life after intensive care. This is a single center randomised controled study comprising patients ≥45 years of age staying 5 days or more in the intensive care unit (ICU). The design is factorial. Inclusion takes place when the patient is leaving the ICU.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients ≥45 years with LOS ≥ 5days

Exclusion Criteria:

* Patients < 45 years, Cerebral function that make cooperation impossible, Fractures in the spine, pelvis and/or lower extremities, Unable to perform the intervention LOS < 5 days

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-02 (Estimated); Primary Completion 2016-02 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
6 minutes walking test (6MWT) (when the patient leave hospital, 12 weeks and 12 months) | One year

SECONDARY OUTCOMES:
Isometric quadriceps strength, Isometrisk handgrip strength, Bodyweight Bodycomposition (Dexa) | One year

OTHER OUTCOMES:
Quality of life SF-36 (when leaving hospital, after 12 weeks and 12 months Body weight (leaving the ICU, after 12 weeks, after 12 months) Body composition (leaving the ICU, after 12 weeks, after 12 months) | One year